CLINICAL TRIAL: NCT04341675
Title: Sirolimus Treatment in Hospitalized Patients With COVID-19 Pneumonia (The SCOPE Trial)
Brief Title: Sirolimus Treatment in Hospitalized Patients With COVID-19 Pneumonia
Acronym: SCOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Nishant Gupta, MD, MS, Adjunct Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-0337
Record Dates: First submitted 2020-04-05; First posted 2020-04-10 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Randmized, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sirolimus (Active Comparator): Sirolimus 6mg on day 1 followed by 2mg daily for the next 13 days or until hospital discharge, whatever happens sooner.
  Interventions: Drug: Sirolimus
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — Sirolimus 6mg daily on Day 1 followed by 2mg daily for the next 13 days for a total treatment duration of 14 days or hospital discharge, whatever happens sooner.
  Other Names: Rapamycin
  Arms: Sirolimus
Drug: Placebo — Matching placebo
  Other Names: placebo capsules
  Arms: Placebo

SUMMARY:
The main objective of our study is to determine if treatment with sirolimus can improve clinical outcomes in hospitalized patients with COVID-19. The investigators will employ a randomized, double blind, placebo-controlled study design. 28 subjects were randomized in a 2:1 fashion to receive sirolimus or placebo. Sirolimus will be given as a 6mg oral loading dose on day 1 followed by 2mg daily for a maximum treatment duration of 14 days or until hospital discharge, whichever happens sooner. Chart reviews will be conducted daily to determine changes in clinical status, concomitant medications and laboratory parameters. Study specific biomarkers will be measured at baseline and then at days 3, 7 and 14.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the trial must meet all of the following criteria.

* Confirmed COVID-19 pneumonia
* Hypoxia as defined by room air oxygen saturation less than 92% or supplemental oxygen requirement
* Presence of at least one additional biomarker that has been shown to predict poor prognosis: a) serum ferritin ≥500ug/l, b) LDH ≥250U/L, c) d-dimer ≥1ug/L, or d) lymphopenia as defined by absolute lymphocyte count <1,000/uL
* Age ≥ 18 years
* Completed informed consent

Exclusion Criteria:

Subjects who meet ANY of the following criteria are not eligible for enrollment as study participants:

* Known allergy or hypersensitivity to sirolimus
* Inability or refusal to provide informed consent
* Advanced respiratory support (high flow oxygen ≥ 15 L/min, CPAP, non-invasive or invasive mechanical ventilation)
* Active enrollment in other interventional clinical drug trials. Co-enrollment in observational studies and biorepositories is allowed.
* Pregnant women
* Breast feeding
* On chronic immunosuppression for other medical conditions such as rheumatological disorders, inflammatory bowel disease, or in patients with organ transplants. A list of these medications is provided in Section 12.3.4
* Any clinically significant medical disease which in the opinion of the investigator precludes the patient from enrolling in the trial, including (but not limited to):

  * History of liver cirrhosis
  * End stage renal disease or need for renal replacement therapy
  * Decompensated heart failure
  * Known active tuberculosis or history of incompletely treated tuberculosis
  * Uncontrolled systemic bacterial or fungal infections
  * Active viral infection other than COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nishant Gupta, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - Loyola University Medical Center, Chicago, Illinois
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Yes Data will be publicly available once the study in published. Deidentified data will be shared with a data use agreement between the requesting entity and the University of Cincinnati.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after the initial study publication.
Access Criteria: Data use agreement between the University of Cincinnati and the requesting entity.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus | Placebo
Started | 18 | 10
Completed | 18 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus | Placebo | Total
Number analyzed (Participants) | 18 | 10 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (15) | 57 (14) | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 15 | 9 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Are Alive and Free From Advanced Respiratory Support Measures at Day 28.
Description: Death or progression to respiratory failure requiring advanced support measures, either due to inadequate ventilation (non-invasive or invasive mechanical ventilation) or inadequate oxygenation (CPAP* or high flow supplemental oxygen at rates ≥ 15 liters/minute), in patients given sirolimus compared to the placebo group.
  * CPAP use for known obstructive sleep apnea will not be considered as disease progression.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 18 | 10
Participants | 15 | 8

2. Secondary Outcome: Percentage of Patients Surviving to Hospital Discharge
Description: Survival to hospital discharge
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 18 | 10
Participants | 17 | 9

3. Secondary Outcome: Drug Safety Profile
Description: Number of patients with adverse events
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 18 | 10
Participants | 9 | 5

4. Secondary Outcome: Duration of Hospital Stay
Description: Length of hospitalization is measured as the number of days in the hospital from the date of randomization until the date of discharge or death from any cause, whichever came first, assessed up to 28 days post discharge.
Time Frame: days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 18 | 10
days | 9.9 (12.2) | 12.9 (11)

5. Secondary Outcome: Number of Patients Who Require Initiation of Off-label Therapies
Description: Patients needing off-label treatments such as Anti-IL-6 inhibitors at the discretion of primary clinicians
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 18 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Sirolimus | Placebo
All-Cause Mortality (participants affected / at risk) | 1/18 | 1/10
Serious Adverse Events (participants affected / at risk) | 3/18 | 2/10
Other Adverse Events (participants affected / at risk) | 9/18 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=18) | Placebo (N=10)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Need for advanced respiratory support (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=18) | Placebo (N=10)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Thromboembolism (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated liver function tests (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Fluid overload (Cardiac disorders) | 1 (1) | 0 (0)
Abnormal serum electrolytes (Investigations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04341675/Prot_SAP_ICF_000.pdf